CLINICAL TRIAL: NCT04657185
Title: Reducing Perioperative S. Aureus Transmission Via Use of an Evidence-Based, Multimodal Program Driven by an Innovative Software Platform (OR PathTrac)
Brief Title: Reducing Perioperative S. Aureus Transmission Via OR PathTrac
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Collaborators: RDB Bioinformatics (Industry); University of Iowa (Other); Trustees of Dartmouth College (Other)
Responsible Party: Sponsor
Other Study IDs: 00000375
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: S. Aureus Transmission; Surgical Site Infection
Keywords: transmission; surgical site infection; s. aureus
MeSH Terms: conditions — Surgical Wound Infection; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — S. aureus pathogens collected were assigned a unique identification number and stored for future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before OR PathTrac Feedback: Patients undergoing surgery with an evidence-based, multifaceted, perioperative infection control program in place but without OR PathTrac feedback optimization.
- After OR PathTrac Feedback: Patients undergoing surgery with an evidence-based, multifaceted, perioperative infection control program in place AND OR PathTrac feedback optimization.
  Interventions: Other: OR PathTrac Feedback Optimization

INTERVENTIONS:
Other: OR PathTrac Feedback Optimization — OR PathTrac (RDB Bioinformatics, Omaha, NE 68154) uses a systematic phenotypic approach leveraging temporal association to monitor 13 anesthesia work area reservoirs proven to be associated with high-risk intraoperative bacterial transmission events and subsequent infection development.
  Groups: After OR PathTrac Feedback

SUMMARY:
Healthcare-associated infections (HAIs) occur frequently and are associated with patient harm. It is important that healthcare facilities take the necessary steps to prevent the spread of resistant bacteria. ESKAPE bacteria (Enterococcus, S. aureus, Klebsiella, Acinetobacter, Pseudomonas, and Enterobacter spp.) are particularly pathogenic. Isolation of these pathogens from intraoperative reservoirs has been associated with postoperative infection development (i.e. surgical site infections). This project involves implementation of a software platform and bacterial collection system (OR PathTrac) that leverages the epidemiology of intraoperative bacterial transmission to guide dynamic, prospective improvements in perioperative infection control measures. The investigators will assess the effectiveness of OR PathTrac feedback in optimizing an evidence-based, multifaceted, perioperative infection control program.

DETAILED DESCRIPTION:
Our objective was to analyze the impact of surveillance feedback optimization of a multifaceted, perioperative infection control program on S. aureus transmission and SSIs. A multifaceted infection control program was implemented over 8 months (November 2018 to June 2019). A prospective cohort impact study was then conducted over 8 months (July 2019 to March 2020) to compare the incidence of within-case S. aureus transmission (primary outcome) and surgical site infection (secondary outcome) before (4.5 months) and after (3.5 months) implementation of surveillance feedback.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients requiring anesthesia and intravenous catheter placement.

Exclusion Criteria:

* Pediatric patients, without requirement of anesthesia and/or intravenous catheter placement.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing surgery requiring anesthesia and intravascular access.
Sampling Method: Non-Probability Sample
Enrollment: 804 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
within-case S. aureus transmission | From patient entry into the operating room until case end, up to 6 hours
  S. aureus transmission events detected within a surgical case

SECONDARY OUTCOMES:
surgical site infection | Up to 90 days following surgery
  evidence of infection (office note documentation with anti-infective order and/or isolation of one or more potentially pathogenic organisms

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University, Georgetown, District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Other researchers must submit a research proposal to be reviewed by Dr. Wall for determination of release.
Supporting Information: CSR
Time Frame: One year after publication the data will become available and will remain available for one year.
Access Criteria: Submission of a research proposal to be reviewed by Dr. Wall.